CLINICAL TRIAL: NCT02528383
Title: Trial of Vaginal Estrogen for Urogenital Symptom Relief in Women on Aromatase Inhibitors: Systemic Impact Versus Local Objective Benefits and Quality of Life
Brief Title: Trial of Vaginal Estrogen for Urogenital Symptom Relief in Women on Aromatase Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Tannenbaum (Other)
Collaborators: Connecticut Breast Health Initiative (Other)
Responsible Party: Sponsor-Investigator, Susan Tannenbaum, Associate Professor, UConn Health
Organization: UConn Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-143-3
Record Dates: First submitted 2015-08-11; First posted 2015-08-19 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: Postmenopausal Women on Aromatase Inhibitors; Vagifem
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vagifem (Experimental): Postmenopausal women diagnosed with breast cancer, are currently on an anti-estrogen called an aromatase inhibitor and you have agreed to undergo treatment with Vagifem based on your physician's recommendation.
  Interventions: Behavioral: Vagifem

INTERVENTIONS:
Behavioral: Vagifem — Women participating in the study will undergo clinical assessments, blood work and complete the quality of life questionnaire at baseline, 6 weeks and 12 weeks study time points. The following will be assessed:
  1. Effect of low dose Vagifem, 10ug tablet on vaginal atrophy.
  2. Effect of low dose Vagifem, 10ug tablet on sex hormones and bone health biomarkers.
  3. Impact of treatment on quality of life

SUMMARY:
Vagifem, is the most appropriate medication to treat bladder and vaginal symptoms such as vaginal dryness and urinary discomfort. The purpose of this research study is to see the benefit this three month vaginal estrogen tablet, Vagifem, has on the bladder, vaginal symptoms and health. The investigators also want to monitor whether the bones might be impacted by estrogen or its absence. If there is an effect on bones, it means that some estrogen may be absorbed from the tablet to affect other places in the body. The investigators are hoping to prove this is not the case. The investigators will also be measuring the quality of life of women participating in the study.

DETAILED DESCRIPTION:
Breast cancers are made of different subtypes but by far the most common characteristic is their estrogen receptor positivity. Seventy percent of breast cancers are estrogen receptor positive and therefore responsive to the hormone estrogen, which acts as a stimulus for growth and survival of the cancer. Studies have repeatedly shown that estrogen deprivation results in prevention of breast cancer in high-risk women, and reduced recurrence of the cancer both locally and systemically as well as overall survival improvement in those women. The majority of women with estrogen sensitive breast cancer are placed on anti-estrogen therapy to prevent the cancer from returning. Even in menopause, women have estrogen produced in their bodies. Many parts of a woman's body require estrogen for normal functioning and reducing the amount of estrogen can affect women significantly in different ways. Some women have significant symptoms like vaginal dryness, which may result in painful sexual relations, discomfort, and frequent urinary tract (bladder) infections. Although the investigators goal is to reduce estrogen to prevent breast cancer from returning, quality of life (how women feel) matters during treatment which can last 5-10 years. A major question is: how medications such as Vagifem that are used to treat vaginal symptoms affect the rest of the body?

This question has not been fully answered and is the reason this study is being done. The safest topical estrogen, Vagifem, is a commercially available tablet which is placed in the vagina. Vagifem works well in many women and is considered to be safe. It is used by gynecologists and cancer doctors in this setting all the time. It is not a new product and has been on the market for many years. Its effects on other parts of the body have not been tested. The investigators are poised to help answer this question by hypothesizing the following:

1. It is impossible to know what impact a given estrogen level has in distant sites, the investigators will however measure these to see if estrogen levels rise in the blood when women are treated with vaginal estrogen tablets that are commercially available. The investigators hypothesize that there will not be any elevation in measurable estrogen levels using very sensitive assays.
2. The investigators also propose using a topical vaginal estrogen application (one that is commercially available) while carefully monitoring its' effects locally in the vagina and its possible impact on bone health. The investigators expect women to have improved vaginal exams as well as improvement in overall quality of life with this treatment. It is also expected that there will be no impact on bone turnover by this topical estrogen replacement.

Postmenopausal women on aromatase inhibitors interested in study participation will be asked to participate for a three month period.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment of Urogenital symptoms with Vagifem, as deemed appropriate by the treating physician
2. History of breast cancer stages 0-III
3. Currently being treated with Aromatase Inhibitors (brand not restrictive) for 3 months or longer
4. Postmenopausal women including those with medically induced menopause
5. Urogenital symptoms consistent with vaginal atrophy.
6. Age 18 years or greater
7. Able to participate in informed consent process
8. Able to read/speak English
9. Able to take daily doses of Vitamin D and Calcium

Exclusion Criteria:

1. Abnormal or unexplained uterine bleeding
2. Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes in serum estrogen levels | 12 Weeks
  Changes in serum estrogen levels will be measured up to 12 weeks in post-menopausal women receiving adjuvant aromatase inhibitors during treatment with low dose vaginal estradiol 10 ug tablet, Vagifem.

SECONDARY OUTCOMES:
Quality of Life | 12 Weeks
  Measure changes in bone health biomarkers up to 12 weeks in post-menopausal women receiving adjuvant aromatase inhibitors during treatment with low dose vaginal estradiol 10 ug tablet, Vagifem to evaluate wellness of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tannenbaum, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States